CLINICAL TRIAL: NCT00612378
Title: A Multi-center Acute Efficacy Trial of GFX For Reduction of Glabellar Furrowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Cosmetic Intervention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACI 09-003
Record Dates: First submitted 2008-01-18; First posted 2008-02-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Glabellar Furrowing; Forehead Wrinkles
Keywords: Glabellar Furrowing
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: GFX System

INTERVENTIONS:
Device: GFX System — The GFX system employs minimally invasive technique utilizing bi-polar radio frequency (RF) technology. GFX ablates nerves activating the muscles that cause glabellar furrowing.
  Other Names: Radio Frequency Ablation

SUMMARY:
The purpose of this research study is to evaluate the immediate effectiveness of the GFX™ device in reducing the furrows (deep frown lines) between eyebrows (glabellar region).

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the acute ability of GFX to reduce glabellar furrowing.

Patients who have presented to the investigator for correction of glabellar furrows, as classified per the Rated Numeric Kinetic Line Scale Score for Facial Wrinkles Secondary to Hyperkinetic Function (Note: Class 1 or Higher)7 (Appendix N) are candidates for this study. All patients must consent to the procedure and agree to complete their post treatment evaluation visit.

ELIGIBILITY:
Inclusion Criteria:

* Has no medical contraindication
* Presenting for correction of glabellar furrows, as classified per the Rated Numeric Kinetic Line Scale Score for Facial Wrinkles Secondary to Hyperkinetic Function (Class 1 or Higher) are candidates for this study
* Is at least 18 years of age
* Signs a written informed consent
* Understands and accepts the obligation to present for the scheduled follow-up visit
* Understands that the GFX procedure may not be successful.

Exclusion Criteria:

* Has had an injection of botulinum toxin to the target area within the previous 3 months and still exhibits a positive cosmetic effect to the glabellar furrow
* Has had silicone, fat, collagen or a synthetic material placed in the glabellar region or surgical correction or excision of the glabellar furrows
* Has a known bleeding disorder
* Has received or is anticipated to receive anti-platelets, anti-coagulants thrombolytics or cancer therapy
* Is receiving systemic corticosteroids or anabolic steroids (standard doses of inhaled or nasal corticosteroids are acceptable)
* Has a history of chronic or recurrent infection or compromised immune system
* Has severe allergies manifested by a history of anaphylaxis
* Has known lidocaine hypersensitivity
* Is enrolled in another study
* Is Pregnant
* Has history of keloid formation
* The investigator believes the patient is not a suitable candidate for the GFX procedure, or is not likely to receive cosmetic benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Successful result from the GFX procedure acutely, without adverse effect | 7 to 10 days post procedure

SECONDARY OUTCOMES:
Minimal or transient incidence of minor adverse events | 7 to 10 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: James Newman, M.D., Study Director — Director, Premier Plastic Surgery; Academic - Clinical Assistant Professor, Facial Plastic & Reconstructive Surgery and Otholaryngology - Head & Neck Surgery, Stanford University Medical center/Palo Alto VA
Locations (5):
- United States (5):
  - Premier Plastic Surgery, San Mateo, California
  - Speirs Clinic for Plastic Surgery, Colorado Springs, Colorado
  - Ben Lee, MD, LLC, Englewood, Colorado
  - David M. Knize, MD, Englewood, Colorado
  - Jasin Facial Rejuvenation, Tampa, Florida